CLINICAL TRIAL: NCT02093546
Title: A Translational Companion Protocol to GOG229O: A Randomized Phase II Study With a Safety Lead-In to Assess the Antitumor Efficacy of the MEK Inhibitor Trametinib Alone or in Combination With GSK2141795, an AKT Inhibitor, in Patients With Recurrent or Persistent Endometrial Cancer
Brief Title: Biospecimen Collection in Assessing the Effect of Trametinib With or Without Uprosertib on Biomarkers in Patients With Persistent or Recurrent Endometrial Cancer Enrolled on Trial GOG02290
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2013-1029; NCI-2018-02663 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-1029 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2014-03-17; First posted 2014-03-21 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Recurrent Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-correlative (Biospecimen collection): Patients undergo collection of blood at screening, between days 3 and 5, 28, and 56. Patients also undergo collection of tumor biopsy at screening and day 28.
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and tumor

SUMMARY:
This trial assesses blood and tumor samples for the effect of trametinib with or without uprosertib on biomarkers in patients enrolled on trial GOG02290 with endometrial cancer that is persistent or has come back. Biomarkers found in the blood and tissue may be related to the reaction or response to the study drugs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To explore the impact of trametinib alone or in combination with uprosertib (GSK2141795) on RAF-MEK-ERK and PI3K pathway signaling.

SECONDARY OBJECTIVES:

I. To examine associations with early changes in functional proteomic biomarkers in tumor biopsies before and after treatment and tumor response in two subgroups of patients with recurrent or persistent endometrial cancer who are treated with trametinib alone or in combination with GSK2141795.

II. To examine levels of circulating tumor cells in blood samples before and after treatment and correlate with tumor response in two subgroups of patients with recurrent or persistent endometrial cancer who are treated with trametinib alone or in combination with GSK2141795.

III. To examine the bRaf/cRaf dimer or Raf/KSR/Mek1 dimers in paraffin sections from these patients before treatment by proximity ligation assay (PLA) assays.

IV. To quantify exosomes from these patients before and after treatment by enzyme-linked immunosorbent assay (ELISA) assay with CD63 antibody and explore bRaf/cRaf dimer or Raf/KSR/Mek1 dimers in exosomes from these patients before and after treatment by PLA assays.

OUTLINE:

Patients undergo collection of blood at screening, between days 3 and 5, 28, and 56. Patients also undergo collection of tumor biopsy at screening and day 28.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be enrolled on GOG0229O
* Patients must have tissue available for molecular analysis. This can be tissue obtained at time of current recurrence or archival tissue from primary diagnosis or recurrence
* Patients must have disease lesions that are amenable to pre- and post- treatment biopsy
* Patients must have signed an approved informed consent and authorization permitting release of personal health information

Exclusion Criteria:

* Patients unwilling to undergo a biopsy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MDACC Participants
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2004-08-13 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Change in biomarker expression | Pre-treatment to post-treatment
  Will use descriptive statistics and graphical methods to compare pre-treatment to post-treatment changes in biomarker expression between patients with and without each type of response for each treatment arm and subgroup. Will estimate mean changes from pre-treatment to each post-treatment assessment with 95% confidence intervals. will use a 2-sample t-test to compare treatment arms with respect to the mean change in biomarker expression. Will use a 2-sample Wilcoxon rank sum test to compare treatment arms with respect to the median change in biomarker expression. This testing may also be restricted to specific subgroups (e.g., patients with complete response), depending on the characteristics of patients accrued. Will also use regression methods to model the change in biomarker expression with time and type of response.

SECONDARY OUTCOMES:
Circulating tumor cells (CTCs) levels | Up to 15 years
  Will use descriptive statistics and graphical methods to compare the numbers of circulating tumor cells (CTCs) over time for patients with and without each type of response for each treatment arm and subgroup. Will estimate with 95% confidence intervals the mean number of CTCs at each assessment time for patients with and without each type of response for each treatment arm and subgroup.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Westin, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org